CLINICAL TRIAL: NCT02935829
Title: Short-term Effects of a Low Glycemic Index Snack Including Carob on Postprandial Glycemic Responses, Energy Intake and Satiety in Normal-weight, Healthy Adults
Brief Title: Short-term Effects of a Carob Snack on Postprandial Glycemic Responses and Energy Intake and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Lecturer in Nutrition and Metabolism, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 304
Record Dates: First submitted 2016-05-24; First posted 2016-10-18 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetite; Lack or Loss, Nonorganic Origin
Keywords: energy intake; blood glucose; carob flour
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Glucose as reference food (Experimental): Ten healthy, normal-weight subjects (male: 6, female: 4) after 10-14 hr fast, consumed 25g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from carob snack and chocolate cookie, one time, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food
- Carob preload (Experimental): Fifty healthy subjects (male: 22, female: 28) were offered a standardized breakfast and 2h after consumed one of the two preloads (carob snack and chocolate cookie) served as snack in random order. Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). Foods were weighed at the time of serving and any leftovers were weighed again after meal to determine the amount of food consumed. Fingertip capillary blood glucose samples were collected before and after foods. Subjective appetite ratings were collected using 100mm visual analogue scales (VAS).
  Interventions: Other: Carob preload
- White bread as reference food (Experimental): Ten healthy, normal-weight subjects (male: 6, female: 4) after 10-14 hr fast, consumed 25g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from carob snack and chocolate cookie, one time, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: White bread as reference food
- Carob snack as test food (Experimental): Ten healthy, normal-weight subjects (male: 6, female: 4) after 10-14 hr fast, consumed 25g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from carob snack and chocolate cookie, one time, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Carob snack as test food
- Chocolate cookie snack as test food (Experimental): Ten healthy, normal-weight subjects (male: 6, female: 4) after 10-14 hr fast, consumed 25g available carbohydrate from white bread and glucose, two times, in different weeks as reference foods along with 250ml water; and 25g available carbohydrates from carob snack and chocolate cookie, one time, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Chocolate cookie snack as test food
- Chocolate cookie preload (Experimental): Fifty healthy subjects (male: 22, female: 28) were offered a standardized breakfast and 2h after consumed one of the two preloads (carob snack and chocolate cookie) served as snack in random order. Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). Foods were weighed at the time of serving and any leftovers were weighed again after meal to determine the amount of food consumed. Fingertip capillary blood glucose samples were collected before and after foods. Subjective appetite ratings were collected using 100mm visual analogue scales (VAS).
  Interventions: Other: Chocolate cookie preload

INTERVENTIONS:
Other: Glucose as reference food — Ten subjects (male: 6, female: 4) consumed 25g glucose diluted in 250ml water, two times, in different weeks, within 5-10 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Glucose as reference food
Other: White bread as reference food — Ten subjects (male: 6, female: 4) consumed 25g available carbohydrate from white bread along with 250ml water, two times, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: White bread as reference food
Other: Carob snack as test food — Ten subjects (male: 6, female: 4) consumed 25g available carbohydrate from carob snack along with 250ml water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Carob snack as test food
Other: Chocolate cookie snack as test food — Ten subjects (male: 6, female: 4) consumed 25g available carbohydrate from chocolate cookie snack along with 250ml water, one time, in different weeks, within 10-15 min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120 min.
  Arms: Chocolate cookie snack as test food
Other: Carob preload — Fifty healthy subjects (male: 22, female: 28) consumed a standardized breakfast (bread and honey) and 2h after were offered a preload given as snack (40g carob snack). Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). The meal consisted of rice, roasted chicken breast and chocolate cake. Foods were weighed before serving and any leftovers were weighed again after meal. Fingertip capillary blood glucose samples were taken before breakfast, 120min after breakfast; before preload, 120minand 180minpost-preload consumption; before meal (lunch and dessert), 60minand 120min post-meal consumption. Subjective appetite ratings were assessed with 100mm VAS.
  Arms: Carob preload
Other: Chocolate cookie preload — Fifty healthy subjects (male: 22, female: 28) consumed a standardized breakfast (bread and honey) and 2h after were offered a preload given as snack (40g chocolate cookie). Three hours after, subjects were given ad libitum access to a meal (lunch and dessert). The meal consisted of rice, roasted chicken breast and chocolate cake. Foods were weighed before serving and any leftovers were weighed again after meal. Fingertip capillary blood glucose samples were taken before breakfast, 120min after breakfast; before preload, 120minand 180minpost-preload consumption; before meal (lunch and dessert), 60minand 120min post-meal consumption. Subjective appetite ratings were assessed with 100mm VAS.
  Arms: Chocolate cookie preload

SUMMARY:
This study investigated any potential associations between two preloads offered as snacks and postprandial glycemic response, subjective and objective appetite and energy intake in healthy, normal-weight adults.

DETAILED DESCRIPTION:
This study aimed at 1. firstly determine the glycemic index (GI) of a carob snack compared with an isoenergetic, equal weight chocolate cookie and 2. test the hypothesis that a carob preload consumed as snack before a meal, compared to chocolate cookie would: (a) have greater short-term effect on satiety measured by subsequent ad libitum meal intake, (b) induce greater satiety as assessed by visual analogue scales (VAS), and (c) reduce postprandial glycemic response.

ELIGIBILITY:
Inclusion Criteria:

- Healthy, non-smoking, non-diabetic men and women individuals with normal body mass index (BMI; between 18.5 and 24.9 kg/m2)

Exclusion Criteria:

* Severe chronic disease (e.g. tumors, manifest coronary heart disease, diabetes mellitus, severe kidney or liver conditions, endocrine and immunological conditions)
* Gastrointestinal disorders (e.g. chronic inflammatory bowel disease)
* Lactose intolerance
* Pregnancy
* Competitive sports
* Lactation
* Alcohol
* Drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose and subjective appetite ratings | 7 hours
  Clinically useful change in serum glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test. Useful change in subjective appetite (hunger, desire to eat, motivation to eat, preoccupation with thoughts of food, thirst) scores from 100mm VAS

SECONDARY OUTCOMES:
Subjective appetite ratings | 6 hours
  Useful change in subjective appetite (hunger, desire to eat, motivation to eat, preoccupation with thoughts of food, thirst) scores from 100mm VAS
Energy intake after preload | 2 hours
  Useful change in energy intake the day of the intervention (actual weighing of foods consumed and leftovers and 24hr recall)
Energy intake next 24hours | 2 days
  Useful change in energy intake in the next 24hr (24hr recall) after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No